CLINICAL TRIAL: NCT04556877
Title: Investigation of the Effects of Different Intra-abdominal Pressures on Optic Nerve Size Measured by Orbital USG in Patients Undergoing Major Abdominal Surgery
Brief Title: Different Intra-abdominal Pressures and Optic Nerve Size
Status: Completed | Type: Observational
Sponsor: Trakya University (Other)
Responsible Party: Principal Investigator, Prof Mehmet Turan Inal, Prof, Trakya University
Other Study IDs: TUTF 2018/230
Record Dates: First submitted 2020-09-07; First posted 2020-09-21 (Actual); Last update posted 2020-09-21 (Actual); Status verified 2020-09

CONDITIONS: Major Surgery; Intraabdominal Hypertension; Optic Nerve Congestion
MeSH Terms: conditions — Intra-Abdominal Hypertension

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Intraabdominal pressure under 12 mmHg: Patients with intraabdominal pressure under 12 mmHg
  Interventions: Procedure: Intraabdominal pressure and optic nerve diameters
- Intraabdominal pressure between 12-20 mmHg: Patients with intraabdominal pressure between 12-20 mmHg
  Interventions: Procedure: Intraabdominal pressure and optic nerve diameters
- Intraabdominal pressure over 20 mmHg: Patients with intraabdominal pressure over 20 mmHg
  Interventions: Procedure: Intraabdominal pressure and optic nerve diameters

INTERVENTIONS:
Procedure: Intraabdominal pressure and optic nerve diameters — Measuring Intraabdominal pressure with a Foley cathater and measuring optic nerve diameters with a USG

SUMMARY:
In intensive care patients, high intraabdominal pressure is frequently encountered. Intra-abdominal pressure is often measured as high, especially after major abdominal surgery procedures. In recent years, various studies have reported that the increase in optic nerve diameter measured by ultrasound correlates with the level of intracranial pressure. Optic nerve diameter measurement with ultrasound is a non-invasive procedure. Intra-abdominal pressure measurements are also routinely performed in intensive care patients. In the measurement of abdominal pressure, the bladder catheter, which is already available in every patient who comes to intensive care, is used. In this study, the intra-abdominal pressure values present in the file of each patient undergoing major abdominal surgery who were taken to intensive care unit will be taken. Orbital USG will be performed on the 6th, 12th and 24th hours on admission to the intensive care unit to measure the diameter of the optic nerve, and the relationship between the intra-abdominal pressure value and optic nerve diameters will be investigated.

DETAILED DESCRIPTION:
In intensive care patients, high intraabdominal pressure is frequently encountered. Intra-abdominal pressure is often measured as high, especially after major abdominal surgery procedures. This situation creates ischemia in the abdominal organs in the patient, decreases venous return as a result of inferior vena cava compression and leads to a decrease in cardiac output. In addition, intracranial pressure frequently increases as a result of the venous circulation being affected. In recent years, various studies have reported that the increase in optic nerve diameter measured by ultrasound correlates with the level of intracranial pressure. Optic nerve diameter measurement with ultrasound is a non-invasive procedure. Intra-abdominal pressure measurements are also routinely performed in intensive care patients. In the measurement of abdominal pressure, the bladder catheter, which is already available in every patient who comes to intensive care, is used. In this study, the intra-abdominal pressure values present in the file of each patient undergoing major abdominal surgery who were taken to intensive care unit will be taken. Orbital USG will be performed on the 6th, 12th and 24th hours on admission to the intensive care unit to measure the diameter of the optic nerve, and the relationship between the intra-abdominal pressure value and optic nerve diameters will be investigated.

ELIGIBILITY:
Inclusion Criteria:

Having had major abdominal surgery

Exclusion Criteria:

1. pregnant patients
2. Patients whose bladder catheter cannot be inserted
3. Patients with diagnosed or suspected brain death

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Postoperative patients followed in intensive care
Sampling Method: Non-Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2018-06-15 (Actual); Primary Completion 2020-06-15 (Actual); Study Completion 2020-06-15 (Actual)

PRIMARY OUTCOMES:
optic nerve diameter | within 2 hours of admission
  measuring optic nerve diameter
optic nerve diameter | at 6.hour
  measuring optic nerve diameter
optic nerve diameter | at 12.hour
  measuring optic nerve diameter
optic nerve diameter | at 24.hour
  measuring optic nerve diameter

CONTACTS AND LOCATIONS:
Locations (1):
- Trakya University, Edirne, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided